CLINICAL TRIAL: NCT00765479
Title: Randomized Placebo-Controlled Adjuvant Study of Prevention of Prostate Cancer Recurrence After Radical Prostatectomy by Soy Protein Isolate
Brief Title: Soy Protein in Preventing Recurrent Cancer in Patients Who Have Undergone Surgery for Stage II Prostate Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000615902; UIC-2006-0706
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-08

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Soybean Proteins

ARMS (2):
- Arm I (Experimental): Patients receive an oral soy protein isolate beverage once daily.
  Interventions: Dietary Supplement: soy protein isolate
- Arm II (Placebo Comparator): Patients receive an oral casein placebo beverage once daily.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: soy protein isolate — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Soy protein may help prevent prostate cancer recurrence in patients who have undergone surgery for prostate cancer.

PURPOSE: This randomized phase II/III trial is studying how well soy protein works and compares it to a placebo in preventing recurrent cancer in patients who have undergone surgery for stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether soy protein isolate reduces the PSA failure rate and time to PSA failure within 2 years following radical prostatectomy in patients who are at high risk for prostate cancer recurrence.
* Determine the effects of soy protein isolate on intermediate biomarkers of steroid hormone axis (testosterone, estradiol, and SHBG) and thyroid activity (T3 and T4).
* Determine the effects of soy protein isolate on intermediate biomarkers of apoptosis (soluble Fas and Fas-ligand), angiogenesis (VEGF and bFGF), antioxidant activity (8-isoprostanes), and IGF axis (IGF-1 and IGFBP-3).
* Compare patients who are equol producers to those who are non-producers.

OUTLINE: This is a multicenter study. Patients are stratified according to hospital/clinic site (NYU vs UIC or Jesse Brown VA Medical Center vs other sites), number of high-risk characteristics (1 vs > 1), and race (African American vs non-African American [i.e., non-Hispanic White, Hispanic, Asian, and other]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive an oral soy protein isolate beverage once daily.
* Arm II: Patients receive an oral casein placebo beverage once daily. Treatment in both arms continues for up to 2 years in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for biomarker laboratory studies. Samples are analyzed to measure PSA levels by Tosoh PSA assay; cholesterol levels; isoflavone and equol concentrations by HPLC and ESA; and indicators of steroid hormone axis (testosterone, estradiol, and SHBG), indicators of thyroid activity (T3 and T4), indicators of apoptosis (soluble Fas and Fas-ligand), indicators of angiogenesis (VEGF and bFGF), indicators of oxidative stress (8-isoprostanes), and indicators of IGF axis (IGF-1 and IGFBP-3) by ELISA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate cancer

  * Clinically localized (T1c or T2) disease
* At high risk for recurrence, as defined by ≥ 1 of the following:

  * Preoperative PSA > 20.0 ng/mL
  * Seminal vesicle invasion
  * Extracapsular extension (excluding the bladder neck)
  * Positive surgical margins (excluding apical margins)
  * Micrometastases in any removed pelvic lymph nodes
  * Final Gleason score of ≥ 8
* Must have undergone radical prostatectomy for prostate cancer within the past 4 months
* Must have an undetectable PSA (< 0.07 ng/mL) at baseline, as measured by Tosoh PSA assay
* No clinical evidence of locally recurrent or metastatic disease

PATIENT CHARACTERISTICS:

* No significant intake of soy (i.e., more than once a week) at baseline including, but not limited to, any of the following:

  * Vegetarians who regularly consume soy products (e.g., tofu)
  * Individuals with customary Asian dietary habits, including regular intake of soy products
  * Individuals who use soy-based milk replacements
* No anemia, iron deficiency problems, or subclinical iron deficiency at baseline
* No diabetes
* No thyroid disease
* No requirement for a sodium-free diet
* No substantive tendency to be constipated (i.e., ≥ grade 2 constipation experienced regularly)
* No medical problem that would preclude the consumption of the soy containing beverage powder, including allergies against soy (or milk protein)
* No concurrent major disease, including major mental disease or major substance abuse problems
* No significant side effects from medication

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent radiotherapy or hormonal therapy
* No other concurrent adjuvant therapy for prostate cancer

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2006-12; Primary Completion 2011-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Two-year PSA failure rate (as surrogate for recurrence)
Time to PSA failure

SECONDARY OUTCOMES:
Isoflavone uptake or compliance as measured by serum isoflavone concentration
Serum total cholesterol levels
Steroid hormone axis as measured by serum testosterone, estradiol, and SHBG levels
Thyroid activity as measured by serum T3 and T4 levels
Apoptotic activity as measured by serum soluble Fas and Fas-ligand levels
Angiogenesis as measured by serum VEGF and bFGF levels
Oxidative stress as measured by serum 8-isoprostane levels
IGF axis as measured by serum IGF-1 and IGFBP-3 levels
Equol production as measured by serum equol concentration

CONTACTS AND LOCATIONS:
Overall Officials: Maarten C. Bosland, DVSc, PhD, Principal Investigator — University of Illinois at Chicago; Roohollah Sharifi, MD — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Bosland MC, Enk E, Schmoll J, Schlicht MJ, Randolph C, Deaton RJ, Xie H, Zeleniuch-Jacquotte A, Kato I. Soy protein supplementation in men following radical prostatectomy: a 2-year randomized, placebo-controlled clinical trial. Am J Clin Nutr. 2021 Apr 6;113(4):821-831. doi: 10.1093/ajcn/nqaa390. PMID 33564828
- [Derived] Bosland MC, Huang J, Schlicht MJ, Enk E, Xie H, Kato I. Impact of 18-Month Soy Protein Supplementation on Steroid Hormones and Serum Biomarkers of Angiogenesis, Apoptosis, and the Growth Hormone/IGF-1 Axis: Results of a Randomized, Placebo-Controlled Trial in Males Following Prostatectomy. Nutr Cancer. 2022;74(1):110-121. doi: 10.1080/01635581.2020.1870706. Epub 2021 Jan 12. PMID 33432829
- [Derived] Bosland MC, Kato I, Zeleniuch-Jacquotte A, Schmoll J, Enk Rueter E, Melamed J, Kong MX, Macias V, Kajdacsy-Balla A, Lumey LH, Xie H, Gao W, Walden P, Lepor H, Taneja SS, Randolph C, Schlicht MJ, Meserve-Watanabe H, Deaton RJ, Davies JA. Effect of soy protein isolate supplementation on biochemical recurrence of prostate cancer after radical prostatectomy: a randomized trial. JAMA. 2013 Jul 10;310(2):170-8. doi: 10.1001/jama.2013.7842. PMID 23839751